CLINICAL TRIAL: NCT00050102
Title: A Randomized Study Comparing MDX-010 (CTLA-4) Alone or in Combination With DTIC in the Treatment of Patients With Chemotherapy Naїve Metastatic Melanoma.
Brief Title: Comparison Study of MDX-010 (CTLA-4) Alone and Combined With DTIC in the Treatment of Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDX010-08; CA184-013 (Other: BMS)
Record Dates: First submitted 2002-11-21; First posted 2002-11-22 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen

INTERVENTIONS:
Drug: MDX-010 (CTLA-4)

SUMMARY:
The objectives of this study are to determine the safety and activity profile of multiple doses of MDX-010, and to determine the whether the addition of cytotoxic chemotherapy (decarbazine [DTIC]) can augment the effects of MDX-010 in patients with chemotherapy naïve metastatic melanoma with a tolerable toxicity profile.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of unresectable metastatic melanoma.
* No prior chemotherapy for melanoma, and no chemotherapy for other malignancies within 5 years and at least 4 weeks since treatment (surgery, radiation, or immunotherapy) for melanoma.

Exclusion Criteria

Patients who exhibit any of the following conditions at screening will not be eligible for admission into the study:

* Any other prior malignancy, except for the following: adequately treated basal or squamous cell skin cancer or superficial bladder cancer, or any other cancer from which the patient has been disease-free for >=5 years.
* Active autoimmune disease.
* Active infection requiring therapy, or chronic active HBV or HCV, or confirmed reactivity with HIV tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (9):
  - Arizona Cancer Center, Tucson, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Northern California Melanoma Center, San Francisco, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Indiana Oncology/ Hematology Consultants, Indianapolis, Indiana
  - Piedmont Oncology Specialists, Charlotte, North Carolina
  - Joe Arrington Cancer. Research & Treatment Center, Lubbock, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Hersh EM, O'Day SJ, Powderly J, Khan KD, Pavlick AC, Cranmer LD, Samlowski WE, Nichol GM, Yellin MJ, Weber JS. A phase II multicenter study of ipilimumab with or without dacarbazine in chemotherapy-naive patients with advanced melanoma. Invest New Drugs. 2011 Jun;29(3):489-98. doi: 10.1007/s10637-009-9376-8. Epub 2010 Jan 16. PMID 20082117